CLINICAL TRIAL: NCT06544707
Title: A Phase 3b Open-Label Study Designed to Evaluate Tear Production Stimulated by 0.003% AR-15512
Brief Title: A Study Designed to Evaluate Tear Production
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEF512-E002
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease
Keywords: Dry Eyes; Eye Drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.003% AR-15512 (Experimental): One drop of 0.003% AR-15512 ophthalmic solution in each eye in a staggered cadence (left eye followed by dosing of the right eye, separated by approximately 2-4 hours)
  Interventions: Drug: 0.003% AR-15512 ophthalmic solution

INTERVENTIONS:
Drug: 0.003% AR-15512 ophthalmic solution — Investigational ophthalmic solution administered via topical instillation
  Other Names: TRYPTYR®; Acoltremon ophthalmic solution 0.003%

SUMMARY:
The purpose of this study is to evaluate tear production following acute administration of AR-15512 ophthalmic solution 0.003% (0.003% AR-15512) in subjects with dry eye disease (DED).

DETAILED DESCRIPTION:
Qualified subjects will attend a single visit.

This is a Phase 3b, 2-stage study. In Stage 1, approximately 40 subjects will be enrolled, after which the study will be paused and an interim analysis will be conducted. Results from the Stage 1 analysis will help inform the design of Stage 2. An additional 40 subjects are planned for Stage 2.

For both stages, the primary endpoint and analysis will remain the same. Stage 2 will be tested independently with no pooling of data between stages.

ELIGIBILITY:
Key Inclusion Criteria:

* Within the last 12 months, have a previous history of dry eye disease, either clinician diagnosed or patient reported.
* Within the last 6 months, have used, or desired to use artificial tears for dry eye symptoms.
* Corrected visual acuity score of 20/200 or better in both eyes.
* Good general and ocular health, as determined by the investigator using medical history, ophthalmic examination and history.
* Other protocol specified inclusion criteria may apply.

Key Exclusion Criteria:

* Current evidence of any clinically significant ophthalmic disease other than dry eye (for example, glaucoma or macular degeneration).
* History of ocular surgery within 1 year of the Study Visit.
* Use of contact lenses in either eye within 7 days of the Study Visit.
* Use of lid hygiene (all forms of lid care) or heat masks within 7 days of the Study Visit.
* Use of any topical ocular anti-inflammatory medications, any topical ocular corticosteroid, or any non-steroidal-anti-inflammatory agents within 30 days of the Study Visit.
* Used artificial tears within 2 hours of the Study Visit.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 investigative site located in the United States.
Pre-assignment Details: This reporting group includes all subjects treated with 0.003% AR-15512 (81).
Groups:
- 0.003% AR-15512 - Stage 1; 0.003% AR-15512 - Stage 2: One drop of 0.003% AR-15512 ophthalmic solution in each eye in a staggered cadence (left eye followed by dosing of the right eye, separated by approximately 2-4 hours)
Period: Overall Study
Arm/Group | 0.003% AR-15512 - Stage 1 | 0.003% AR-15512 - Stage 2
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All subjects who have received at least one dose of 0.003% AR-15512 and have pre-drop and 3-minute post-drop tear meniscus height measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.003% AR-15512 - Stage 1 | 0.003% AR-15512 - Stage 2 | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.83) | 62.5 (14.80) | 61.5 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 30 | 30 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 9 | 18
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 31 | 28 | 59
  Multi-Racial | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Tear Meniscus Height (TMH) at Minute 3 - Stage 1
Description: TMH (the distance between the line of reflection along the top of the tear prism to the edge of the central lower eyelid) was measured pre-instillation and post-instillation in micrometers using optical coherence tomography (OCT), a non-invasive imaging test that uses light waves to take cross-section pictures of the eye. A normal TMH range falls between 200 and 400 micrometers. Measurements below this range may indicate dry eye disease. A positive change value indicates an improvement. One eye (study eye, defined as the left eye) contributed data to the analysis.
Time Frame: Day 1, Minute 0 pre-instillation (Baseline); Day 1, Minute 3 post-instillation
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 - Stage 1
Number analyzed (Participants) | 40
Number analyzed (eyes) | 40
micrometers | 519.65 (515.561)
Statistical Analysis 1: Comparison: 0.003% AR-15512 - Stage 1; Test type: Other — Single-arm study; p < 0.0001, t-test, 1 sided — P-value one-sided significance level = 5%

2. Primary Outcome: Mean Change From Baseline in Tear Meniscus Height (TMH) at Minute 3 - Stage 2
Description: as for outcome 1
Time Frame: Day 1, Minute 0 pre-instillation (Baseline); Day 1, Minute 3 post-instillation
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 - Stage 2
Number analyzed (Participants) | 41
Number analyzed (eyes) | 41
micrometers | 503.80 (559.552)
Statistical Analysis 1: Comparison: 0.003% AR-15512 - Stage 2; Test type: Other — Single arm study; p < 0.0001, t-test, 1 sided — P-value one-sided significance level = 5%

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent until study exit, approximately 1 day.
Description: An AE was defined as any untoward medical occurrence associated with the administration of the study intervention in humans, whether or not considered to be related to the study intervention. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. The safety analysis set included all subjects who have received at least one dose of 0.003% AR-15512.
Groups:
- Pretreatment: AEs occurring from time of consent until initiation of treatment with 0.003% AR-15512
Arm/Group | Pretreatment | 0.003% AR-15512 - Stage 1 | 0.003% AR-15512 - Stage 2
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/81 | 19/40 | 16/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=81) | 0.003% AR-15512 - Stage 1 (N=40) | 0.003% AR-15512 - Stage 2 (N=41)
Instillation site irritation (General disorders) | 0 (0) | 19 (19) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT06544707/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT06544707/SAP_001.pdf